CLINICAL TRIAL: NCT06950710
Title: Mechanisms of Macrophage Polarization in Hepatic Ischemia-Reperfusion Injury in Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: Mechanisms of Macrophage Polarization in HIRI in Patients With NAFLD
Status: Active, not recruiting | Type: Observational
Sponsor: Zhifeng Gao (Other)
Responsible Party: Sponsor-Investigator, Zhifeng Gao, Chief Physician, Beijing Tsinghua Chang Gung Hospital
Organization: Beijing Tsinghua Chang Gung Hospital (Other)
Other Study IDs: 25304-4-01
Record Dates: First submitted 2025-04-21; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Ischemia-reperfusion Injury; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NAFLD group
  Interventions: Other: NAFLD
- Control group

INTERVENTIONS:
Other: NAFLD — This study is an observational one with no intervention
  Other Names: Control
  Groups: NAFLD group

SUMMARY:
To better understand the occurrence of hepatic ischemia-reperfusion injury (IRI) in patients with non-alcoholic fatty liver disease (NAFLD) and the role of macrophage polarization in this process, this study will retrospectively collect clinical data from patients who underwent partial hepatectomy at Beijing Tsinghua Changgung Hospital between September 2021 and March 2025. Additionally, clinical information and liver blood samples from patients scheduled for partial hepatectomy from April 2025 onward will be prospectively collected. These samples will include normal liver tissue from the resected portion, as well as 5 mL of venous blood obtained before and after surgery. The investigators will compare the severity of hepatic IRI, the expression of macrophage polarization-related proteins, and macrophage polarization markers in blood samples between NAFLD patients and controls. The study aims to determine whether NAFLD patients experience more severe hepatic IRI and to elucidate the role and mechanisms of macrophage polarization in this context. The findings will provide a theoretical basis for understanding the molecular mechanisms underlying hepatic IRI in NAFLD patients, thereby identifying potential therapeutic targets to prevent IRI and improve prognosis in NAFLD patients undergoing partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* The vital organ systems (heart, lungs and kidneys) have sufficient functional reserves.

Exclusion Criteria:

* No hepatic inflow occlusion (Pringle maneuver) was applied during surgery.
* American Society of Anesthesiologists (ASA) Physical Status Classification > Grade III.
* Secondary causes of hepatic steatosis were excluded, including viral hepatitis, drug-induced liver injury, total parenteral nutrition, Wilson's disease, and autoimmune liver diseases.
* Prior chemotherapy or radiotherapy before the planned surgery.
* Use of anticoagulant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing partial hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of transaminase | 7 days after the operation
  ALT、AST

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua Medicine，Tsinghua University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided